CLINICAL TRIAL: NCT04190927
Title: A New Hormone Replacement Paradigm: Physiologic Restoration Using Compounded Biomimetic Estradiol, Progesterone and Testosterone Applied Transdermally in a Rhythmic Dose
Brief Title: A New Hormone Replacement Paradigm: Physiologic Restoration Study
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Women's Hormone Network (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WHN 13/13; 19-71ix (Other: Cottage Hospital Research Institute)
Record Dates: First submitted 2019-11-22; First posted 2019-12-09 (Actual); Last update posted 2020-04-01 (Actual); Status verified 2020-03

CONDITIONS: Menopause; Perimenopausal Disorder; Menopause Related Conditions
Keywords: Menopause; Hormone Replacement Therapy; Bioidentical HRT; Transdermal HRT; Rhythmic Dosing; Physiologic Restoration; Biomimetic HRT

STUDY DESIGN:
Intervention Model Description: Observational, single arm, prospective using a new dosing regimen of an existing biological drug.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Treatment (Experimental): All patients will be symptomatic peri or post menopausal and will all be started on the same protocol. The Dosing schedule of topical estradiol and topical progesterone will be modified for each subject in the first three months to address individual symptoms. The dosing will be relatively unique to each patient. Patients will remain on their dosing schedule for the remainder of the three year study and will be assessed during at the end of the study for changes in mood, symptoms of menopause, breast health, BMD and thickness of uterine lining .
  Interventions: Biological: Compounded topical estradiol and compounded topical progesterone in a carrier cream

INTERVENTIONS:
Biological: Compounded topical estradiol and compounded topical progesterone in a carrier cream — Apply topical compounded estradiol and progesterone in the amount prescribed twice daily for each day of the 28 day lunar or menstrual cycle. Repeat each cycle month. Make note of any AE's so that modifications in dosing can be made.

SUMMARY:
This is a three-year, prospective, observational study looking at the benefits of rhythmically dosed, bio-identical hormones compounded in a carrier cream in 100 symptomatic peri and postmenopausal women. This study will measure changes in cognition, mood, quality of life, endocrine health, bone mineral density, and reduction of the symptoms of menopause and any adverse effects. The objectives of this study are to show that rhythmic dosing of bio-identical hormones that mimic a menstrual cycle, are possible, and may be more beneficial and have fewer side effects than the current standard of care for treating the symptoms of menopause.

DETAILED DESCRIPTION:
"Bio-identical" hormones, which are compounded plant-based hormones synthesized into structurally similar to human estradiol and progesterone molecules, became popular in 2004 by celebrity, Suzanne Somers, who let women know there were natural alternatives to the drugs with hormone-like activity. Compounding hormones makes it easy to make dose adjustments in order to manage symptoms. Using this form of hormone delivery, it is possible to try and replicate a normal physiological reproductive pattern of replacement akin to thyroid replacement, etc. Current short-term studies with bio- identical transdermal estradiol and progesterone have not supported increased breast cancer or other issues such as venous thrombosis7. Even the WHI stated that the increase in breast cancer was due to stimulation of cancers already present.

This study of bio-identical physiologic restoration and dosing of estradiol, testosterone and cyclical transdermal progesterone attempts to replicate the reproductive hormone patterns and levels of a premenopausal woman. This dosing schedule has higher doses and levels than current standard estradiol and progesterone hormone therapy for post menopause women. Research shows that the estradiol peak of a menstrual cycle has an impact on cell signaling and receptor response. For example, TP53, the gene major tumor suppressor gene is under estrogen and progesterone control. At the peaks of estradiol and progesterone, TP53 is up regulated conferring cellular protection against mutations8-14.

Physiologic Restoration (PR) with bio-identical rhythmic dosing was originally developed by S.T. Wiley, who developed a template of hormone doses over time and was meant to be adjusted to the individual women depending on their symptoms and, absorption, metabolism, and response to the program. This study will utilize this concept with some improvements to the original proposed template (Sex, Lies, and Menopause, 2004). This regimen has been in national clinical practice since 2004 and has not been formally studied until now. There is unpublished observational data from Dr. Taguchi's high risk population of oncology patients (Santa Barbara Cottage Hospital IRB# 19-71ix) showing that PR is feasible and manages menopause symptoms well without seemingly more adverse effects and better sense of well being and excellent reversal or improvement of osteoporosis.

ELIGIBILITY:
Inclusion Criteria:

1. Symptomatic perimenopausal or menopausal women as determined by symptoms, history, or labs that confirm menopause status.
2. Any women interested in physiologic restoration for HRT replacement.
3. Women with a history of breast, endometrial or ovarian cancer who are seeking HRT regardless of their diagnosis and recommendations not to have HRT. They must understand the risk and give informed dissent.
4. Hysterectomy.

Exclusion Criteria:

1. Women who are pregnant and or breastfeeding.
2. Women who may be allergic to the base used for compounding.
3. Previous recent (< 12 months) rhythmic dosing hormone protocol.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-06-01 (Estimated); Primary Completion 2023-06-01 (Estimated); Study Completion 2023-08-01 (Estimated)

PRIMARY OUTCOMES:
Change in Symptoms of Menopause | 36 months
  Measure changes in hormone levels and blood chemistry, assess changes in mood and cognitive function, measure changes in brain structure
Compliance of this HRT Regimen | 36 months
  Measure compliance of patients on this specific HRT regimen
Change in Bone Mineral Density | 36 months
  Bone Mineral Density will be monitored for changes

SECONDARY OUTCOMES:
Incidence of adverse effects | 36 months
  Measure incidence of cancer, embolism, coronary artery disease and stroke

CONTACTS AND LOCATIONS:
Overall Officials: Julie Taguchi, MD, Principal Investigator — Principal Investigator

IPD SHARING:
Plan to Share IPD: Yes
After all identifying information is removed from each patient's lab and study results, all results will be made available to the Women's Hormone Network so that they may be used for future study. Each patient will be identified by their last initial and year of birth (e.g. M1950) IPD to be shared are all lab results, blood work, BMD, mammogram, cognitive and mood questionnaires, and MRI, if applicable.
Supporting Information: Study Protocol, CSR
Time Frame: During the study, at years one and two and at the conclusion of the study. Data will be available indefinitely.
Access Criteria: Requests for IPD will be submitted and reviewed by the Women's Hormone Network.

REFERENCES:
- See also: website for the Women's Hormone Network — http://womenshormonenetwork.org